CLINICAL TRIAL: NCT01017055
Title: Voice and Swallowing Outcomes Following Revision Anterior Cervical Spine Surgery
Status: Completed | Type: Observational
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Kirk P. Withrow, MD, Associate Professor of Surgery, University of Alabama at Birmingham
Other Study IDs: IRB-090409003; IRB-090409003 (Other: UAB)
Record Dates: First submitted 2009-11-04; First posted 2009-11-20 (Estimated); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Dysphagia; Dysphonia
MeSH Terms: conditions — Deglutition Disorders; Dysphonia | interventions — Voice

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Voice and Swallowing Evaluations
  Interventions: Other: Voice and Swallowing evaluations

INTERVENTIONS:
Other: Voice and Swallowing evaluations — Fiberoptic exam to evaluate vocal cord and swallowing function

SUMMARY:
Evaluate voice and swallowing outcomes post operatively.

DETAILED DESCRIPTION:
Anterior Cervical Decompression and fusion is one of the most common spinal surgical procedures performed in the United States. Common complications of this type of surgery are difficulty swallowing and nerve dysfunction that can effect voice. The chance of having voice and swallowing disturbances increases if this type of surgery has to be repeated. The purpose of this study is to document the voice and swallowing function of patients undergoing this type of surgery in an effort to find better ways to identify and treat these common complications.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing revision anterior cervical spine surgery

Exclusion Criteria:

* Primary pathology of the upper aero-digestive tract other than mild chronic pharyngitis, pre-existing vocal cord paralysis.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing revision anterior cervical spine surgery
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2009-10-26 (Actual); Primary Completion 2025-12-25 (Actual); Study Completion 2026-01-01 (Actual)

PRIMARY OUTCOMES:
Vocal cord and swallowing function as measured by fiberoptic exam in the otolaryngology clinic pre-op and approximately 3 weeks post op. | 4 weeks

SECONDARY OUTCOMES:
Quality of life as measured by a self-administered 10 point questionnaire. | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: William R Carroll, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- UAB, Birmingham, Alabama, United States